CLINICAL TRIAL: NCT03725800
Title: Rationale and Design of the OCEAN Study (Long-term mOno-antiplatelet Drug Strategy After perCutanEous coronAry interveNtion), A Multicenter, Prospective, Registered Branch of the RESCIND Study
Brief Title: Long-term MOno-Antiplatelet Drug Strategy After PerCutanEous CoronAry InterveNtion
Acronym: RESCIND-OCEAN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); Guangzhou Panyu Central Hospital (Other); First People's Hospital, Shunde China (Other); Second People's Hospital of Foshan City (Unknown); The First People's Hospital of Qingyuan (Unknown); Zhongshan People's Hospital, Guangdong, China (Other); Huadu District People's Hospital of Guangzhou (Other)
Responsible Party: Principal Investigator, Liu yong, MD, PhD, Guangdong Provincial People's Hospital
Other Study IDs: GDREC2018419H
Record Dates: First submitted 2018-10-27; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Antiplatelet Drug-related Gastrointestinal Injury
Keywords: coronary heart disease; mono-antiplatelet drug; antiplatelet-induced gastrointestinal injury symptom; medication adherence; prospective observational study
MeSH Terms: conditions — Coronary Disease; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aspirin: Patients(aged ≥18 years) who have undergone PCI between 1 and 1.5 years, currently alive and is using aspirin for mono-antiplatelet therapy.
- Clopidogrel: Patients(aged ≥18 years) who have undergone PCI between 1 and 1.5 years, currently alive and is using clopidogrel for mono-antiplatelet therapy.
- ASIDE: Patients(aged ≥18 years) who have undergone PCI between 1 and 1.5 years, currently alive and is using ASIDE for mono-antiplatelet therapy.

SUMMARY:
The OCEAN (long-term mOn-antiplatelet drug strategy after perCutanEous coronANy intervention) study is the largest prospective multicenter data base to investigate the long-term incidence and prognosis of the use of agents for antiplatelet-induced GI injury symptoms (AI-GIS) or GI hemorrhage among patients undergoing PCI. The OCEAN study will provide evidence of the long-term incidence and prognosis of use of agents for AI-GIS among patients undergoing PCI. It has the potential to provide an optimal long-term mono-antiplatelet strategy.

DETAILED DESCRIPTION:
This is a multicenter prospective observational study that will collect data on >1000 alive patients who have undergone PCI between 1 and 1.5 years prior at 9 hospitals from October 2018. Adult patients (aged ≥18 years) undergoing PCI and prescribed mono-antiplatelet agents (such as aspirin, dihydroxyaluminum aminoacetate-heavy magnesium carbonate-aspirin, and clopidogrel) are eligible for enrollment. In phase 1, patients will be investigated in a cross-sectional manner for the withdrawal rate of dual antiplatelet agents within 1 year after stent implantation. In phase 2, patients will be followed up at 1, 3, and 6 months for AI-GIS and other outcomes. The primary endpoint is AI-GIS (according to the Gastrointestinal Symptom Rating Scale score) or gastrointestinal hemorrhage. Secondary outcomes will include bleeding, antiplatelet replacement/discontinuation, health economic cost, utilization ratio of gastrointestinal-protective drugs, and MACE.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Currently alive at 1-1.5 years after PCI
3. Considered by the physician to be suitable for long-term treatment with mono-antiplatelet agents and is currently using a mono-antiplatelet drug (aspirin, clopidogrel, or dihydroxyaluminum aminoacetate-heavy magnesium carbonate-aspirin [ASIDE])
4. Provided written informed consent for this study.

Exclusion Criteria:

1. Refusal to sign the informed consent form
2. Acute coronary syndromes
3. Cerebral thrombosis within 1 month or cerebral hemorrhage within 1 year
4. Hematopathy or non-GI bleeding tendency
5. Allergy to aspirin
6. Severe uncontrolled hypertension (>180/110 mmHg)
7. Pregnancy or lactation
8. Drug or alcohol abuse
9. Malignant tumor or <1-year life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OCEAN study is a multicenter, prospective, observational study. The study population will consist of 1000 patients. It will be conducted in 9 centers in China.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Antiplatelet-induced Gastrointestinal Injury Symptom(AI-GIS) | 1 year after PCI
  AI-GIS was estimated according to the Gastrointestinal Symptom Rating Scale(GSRS). This scale included a total of 15 evaluation indicators(Abdominal pains、Heartburn、Acid regurgitation、Sucking sensations in the epigastrium、Nausea and vomiting、Borborygmus、Abdominal distension、Eructation、Increased flatus、Decreased passage of stools、Increased passage of stools、Loose stools、Hard Stools、Urgent need for defecation、Feeling of incomplete evacuation）. The score for each indicator was determined by intensity, frequency, duration, request for relief, and impact on social performance. A score of 0 indicated no or only transient symptoms. A score of 3 indicated continuous discomfort with impact on all social activities. The total minimum score was 0 points and the total maximum score was 45 points. Higher score represented a worse outcome.

SECONDARY OUTCOMES:
Bleeding Events | 1-1.5 years after PCI
  It was estimated according to Thrombolysis in Myocardial Infarction [TIMI] score. This score included two categories: Major bleeding and Minor bleeding. The Major bleeding was defined as: Intracranial or clinically significant overt signs of hemorrhage associated with a greater than 50 g/L decrease in hemoglobin level or an absolute decrease in hematocrit of greater than 15%(when hemoglobin level was not available). The Minor bleeding was defined as: Observed blood loss and a decrease in hemoglobin level of 30 to 50 g/L (or, when hemoglobin level was not available, a decrease in the hematocrit of 9 to 15 percentage points) or a decrease in hemoglobin level of 40 g/L or greater (or ≥12% in hematocrit) if no bleeding site was identifiable. We also monitored for the occurrence of profound thrombocytopenia (<20x103 platelets/μL) or need for transfusion of blood products.
Conversion of Antiplatelet Drug | 1-1.5 years after PCI
  Conversion of antiplatelet drug included brief (1-7 days), temporary (8-30 days), or permanent (>30 days) conversion, according to the continued conversion duration within 1 year after drug-coated stent implantation.
Discontinuation of Antiplatelet Drug | 1-1.5 years after PCI
  Discontinuation of antiplatelet drug included brief (1-7 days), temporary (8-30 days), or permanent (>30 days) discontinuation, according to the continued discontinuation duration within 1 year after drug-coated stent implantation.
Health Economic Costs | 1-1.5 years after PCI
  Health economic costs included the following 3 parts: 1) cost of each of the 3 antiplatelet drugs; 2) cost of each of the 3 antiplatelet drugs plus PPI; and 3) total prescription cost provided at each follow-up time.
Utilization Rate of GI Protection Drug | 1-1.5 years after PCI
  Utilization rate of GI protection drug included brief (1-7 days), temporary (8-30 days), or permanent (>30 days) utilization of PPI, H2RA, sucralfate, or prostaglandins, according to the continued utilization duration within 1 year after drug-coated stent implantation.
Major Adverse Cardiovascular Events | 1-1.5 years after PCI
  All-cause mortality, target vessel revascularization, and non-fatal myocardial infarction (at 3 and 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Liu, MD,PhD, Study Director — Guangdong Cardiovascular Institute,Guangdong General Hospital; Shiqun Chen, MS, Study Director — Guangdong Cardiovascular Institute,Guangdong General Hospital
Locations (7):
- China (7):
  - The First People's Hospital of Shunde, Foshan, Guangdong
  - The Second People's Hospital of Foshan, Foshan, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Huadu District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The First Affiliated Hospital of Clinical Medicine of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong